CLINICAL TRIAL: NCT07106385
Title: The Effectiveness of Repetitive Transcranial Magnetic Stimulation (rTMS) on Improving Sleep Quality in Adults Without Serious Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Cheng Pak Wing, Calvin, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 25-281
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Rtms; Sleep
Keywords: rtms; sleep; health adults
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy adults (Experimental)
  Interventions: Device: rtms

INTERVENTIONS:
Device: rtms — Participants will undergo a treatment protocol involving six sessions of rTMS using the EXOMIND™ device, administered once or twice a week. Each session will deliver 6,300 pulses at alternating frequencies of 12, 15, and 18 Hz, with a total duration of 24 minutes and 30 seconds. The target site would be left dorsolateral prefrontal cortex (DLPFC), determined by the most common used 5-cm rule. The procedure would be conducted in our research centre with medical staff supported.

SUMMARY:
The Effectiveness of Repetitive Transcranial Magnetic Stimulation (rTMS) on

Improving Sleep Quality in Adults Without Serious Mental Illness

Introduction

The investigators would like to invite participants to participate in a study on the efficacy of using magnetic fields to improve sleep quality in adults with no serious mental illness.

The research leader is Dr. Cheng Pak Wing, Assistant Professor, Department of Psychiatry, Queen Mary Hospital/ HKU Li Ka Shing Faculty of Medicine.

Please read the following information carefully. If necessary, participants can discuss with relatives, friends or doctors. If anything is unclear, or if participants would like more information, please ask us. Please carefully consider whether participants are willing to participate in this research.

Research Purpose

Sleep is a fundamental component of overall health and well-being, playing a crucial role in cognitive function, emotional regulation, and physical health. However, sleep complaints are common, even among otherwise healthy adults, often leading to reduced quality of life and increased health risks. The prevalence of poor sleep quality can be attributed to a variety of factors, including stress, lifestyle habits, and environmental disturbances.

rTMS is a non-invasive brain stimulation technique that uses magnetic fields to modulate neural activity in targeted brain regions. Over the years, rTMS has shown promise in treating various mental health conditions, including depression, obsessive-compulsive disorder (OCD) and clinical insomnia.

Research Methods

Participants

Healthy adults aged 18-65 with self-reported sleep complaints.

Treatment protocol

Six sessions of rTMS using the EXOMIND™ device, administered once or twice a week.

Each session will deliver 6,300 pulses at alternating frequencies of 12, 15, and 18 Hz, with a total duration of 24 minutes and 30 seconds.

The target site would be left dorsolateral prefrontal cortex (DLPFC), determined by the most common used 5-cm rule. The procedure would be conducted in the research centre with medical staff supported.

A checklist of potential adverse effects from TMS administration will be referenced from existing literature to monitor tolerability and adverse events during each session. Blood pressure and heart rate will be recorded at the beginning and end of each session.

Assessment

Participants will be assessed at three time points: baseline (pre-intervention), post-intervention, and four weeks post-intervention.

Assessments: Pittsburgh Sleep Quality Index (PSQI), Perceived Stress Scale (PSS), Patient Health Questionnaire-9 (PHQ-9), and home sleep monitoring device.

Demographics: age, gender, years of education, place of birth, marital status, number of children, financial condition, household income, family history of sleep difficulties will be collected upon study entry. Medical history in relation to mental illnesses and medications will also be assessed.

DETAILED DESCRIPTION:
Risks of Participation

Participants may experience mild discomfort from brain stimulation treatment. A small percentage of users may experience dizziness, headache, or nausea. The side effects of brain pulse stimulation therapy are short-lived and are not known to cause any permanent damage. If participants feel unwell after completing the brain pulse stimulation treatment, please inform the staff and therapist.

Note: Patients who have had metal implants in the head, neck, or upper back, or who have had metal teeth/dental trays or pacemakers, should not receive brain stimulation.

Benefits of Participation

The investigators sincerely invite participants to participate in this study.

The valuable information participants provide will help us understand the effect of using magnetic fields to improve sleep quality in adults.

Voluntary Participation

Participation in our research is entirely voluntary and participants have the right to withdraw from research at any time. Participants' decision to participate in or withdraw from the study will not affect participants' existing treatment or services. The information participants provide will be kept strictly confidential and all information will be used for research purposes only.

Financial Costs

Participants will not be charged for the service. Study article will not be continued to be available to subjects after the study until it is commercially available.

Confidentiality of Information

Any information about participants obtained during the research process will be kept strictly confidential. Any information about participants that is released outside the hospital (e.g. in scientific literature or reports) will not have personally identifiable information about participants. Each study participant has the right to access their personal data and publicly reported study results if required, and participants' contact details will be reserved for future follow-up studies.

Personal data will be kept for 5 years after completion of study and publications to keep track on potential side effects related to the intervention. Data will be destroyed after completion of publications.

Under the laws of Hong Kong (especially the Personal Data (Privacy) Ordinance, Cap. 486), participants have the right to keep participants' personal data confidential, such as the collection of personal data in or in connection with this research, Safeguard, retain, manage, control, use (analyze or compare), transfer within or outside Hong Kong, non-disclosure, erasure and/or deal within any way. If participants have any questions, participants can consult the Office of the Privacy Commissioner for Personal Data or call its office (telephone number: 2827 2827) to properly supervise or monitor the protection of participants' personal data so that participants are fully aware and aware of ensuring compliance with the law to protect private data meaning.

By agreeing to participate in this study, participants expressly authorize:

To oversee this study, authorize the principal investigator and his research team and the Institutional Review Board of the University of Hong Kong/ Hospital Authority Hong Kong West Cluster to obtain, use and retain participants in the manner specified in this study and this informed consent, and

Authorize relevant government agencies (such as the Hong Kong Department of Health) to obtain participants' personal data to check and verify the integrity of the research data and assess the consistency of the research agreement with the relevant requirements.

Enquiries

This study has been reviewed and approved by the Institutional Review Board of the University of Hong Kong/ Hospital Authority Hong Kong West Cluster. If participants are willing to participate in the research, please sign the enclosed informed consent form and keep this fact sheet for reference.

The study was coordinated by Dr. Cheng Pak Wing, Assistant Professor, Department of Psychiatry, Faculty of Medicine, The University of Hong Kong.

For enquiries, please contact our Research Assistant at 9016 9487, or Institutional Review Board of the University of Hong Kong/ Hospital Authority Hong Kong West Cluster at 2255 4086.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Aged between 18-65
* Self-reported sleep complaints

Exclusion Criteria:

* Serious mental illness other than primary insomnia
* Severe neurological conditions
* Contraindications for rTMS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2027-06-27 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline: 1-week before rTMS intervention starts Post-intervention: 1-week immediately after the last session of rTMS intervention 4-week post-intervention: 4-week after the last session of rTMS intervention
  Using Pittsburgh Sleep Quality Index (PSQI) to measure subjective sleep quality
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | Baseline: 1-week before rTMS intervention starts Post-intervention: 1-week immediately after the last session of rTMS intervention 4-week post-intervention: 4-week after the last session of rTMS intervention
  Using perceived stress scale (PSS) to evaluate perceived stress levels.
  First, reverse the scores for questions 4, 5, 7, and 8. On these 4 questions, change the scores like this: 0 = 4, 1 = 3, 2 = 2, 3 = 1, 4 = 0.
  * Now add up the scores for each item to get a total. The total score is ___________.
  * Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
    * Scores ranging from 0-13 would be considered low stress.
    * Scores ranging from 14-26 would be considered moderate stress.
    * Scores ranging from 27-40 would be considered high perceived stress
Patient Health Questionnaire-9 (PHQ-9) | Baseline: 1-week before rTMS intervention starts Post-intervention: 1-week immediately after the last session of rTMS intervention 4-week post-intervention: 4-week after the last session of rTMS intervention
  Using Patient Health Questionnaire-9 (PHQ-9) to assess depressive symptoms
  Scoring: add up all checked boxes on PHQ-9 (For every 3 Not at all = 0; Several days = 1; More than half the days = 2; Nearly every day = 3)
  Interpretation of Total Score: Total Score Depression Severity 1-4: Minimal depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20-27: Severe depression
Sleep time and stages | Baseline: 7 consecutive nights before the rTMS intervention starts Post-intervention: 7 consecutive nights after the last session rTMS intervention
  Using sleep watch to measure total sleep time and duration of each sleep stage (in minutes).
  Participants are required to wear a watch when they sleep to monitor their sleep time and duration of each sleep stage. This is to provide an objective data in pre- and post intervention changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, HKU, Hong Kong, Pok Fu Lam, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Protecting participants data

REFERENCES:
- [Background] Voineskos D, Blumberger DM, Rogasch NC, Zomorrodi R, Farzan F, Foussias G, Rajji TK, Daskalakis ZJ. Neurophysiological effects of repetitive transcranial magnetic stimulation (rTMS) in treatment resistant depression. Clin Neurophysiol. 2021 Sep;132(9):2306-2316. doi: 10.1016/j.clinph.2021.05.008. Epub 2021 Jun 1. PMID 34167891
- [Background] Sabe M, Hyde J, Cramer C, Eberhard A, Crippa A, Brunoni AR, Aleman A, Kaiser S, Baldwin DS, Garner M, Sentissi O, Fiedorowicz JG, Brandt V, Cortese S, Solmi M. Transcranial Magnetic Stimulation and Transcranial Direct Current Stimulation Across Mental Disorders: A Systematic Review and Dose-Response Meta-Analysis. JAMA Netw Open. 2024 May 1;7(5):e2412616. doi: 10.1001/jamanetworkopen.2024.12616. PMID 38776083
- [Background] Liang K, Li H, Bu X, Li X, Cao L, Liu J, Gao Y, Li B, Qiu C, Bao W, Zhang S, Hu X, Xing H, Gong Q, Huang X. Efficacy and tolerability of repetitive transcranial magnetic stimulation for the treatment of obsessive-compulsive disorder in adults: a systematic review and network meta-analysis. Transl Psychiatry. 2021 May 28;11(1):332. doi: 10.1038/s41398-021-01453-0. PMID 34050130
- [Background] Zhu L, Dang G, Wu W, Zhou J, Shi X, Su X, Ren H, Pei Z, Lan X, Lian C, Xie P, Guo Y. Functional connectivity changes are correlated with sleep improvement in chronic insomnia patients after rTMS treatment. Front Neurosci. 2023 Apr 17;17:1135995. doi: 10.3389/fnins.2023.1135995. eCollection 2023. PMID 37139515
- [Background] Ma H, Lin J, He J, Lo DHT, Tsang HWH. Effectiveness of TES and rTMS for the Treatment of Insomnia: Meta-Analysis and Meta-Regression of Randomized Sham-Controlled Trials. Front Psychiatry. 2021 Oct 22;12:744475. doi: 10.3389/fpsyt.2021.744475. eCollection 2021. PMID 34744835
- [Background] Sun N, He Y, Wang Z, Zou W, Liu X. The effect of repetitive transcranial magnetic stimulation for insomnia: a systematic review and meta-analysis. Sleep Med. 2021 Jan;77:226-237. doi: 10.1016/j.sleep.2020.05.020. Epub 2020 May 22. PMID 32830052

DOCUMENTS (2):
  • Study Protocol (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT07106385/Prot_000.pdf
  • Informed Consent Form (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT07106385/ICF_001.pdf